CLINICAL TRIAL: NCT01414179
Title: Nutrition Environnement et Santé Cardio Vasculaire NESCAV
Brief Title: NESCAV Nutrition Environment and Cardiovascular Health
Acronym: NESCAV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: CIC-P (Unknown); European Regional Development Fund (Other); Luxembourg Institute of Health (Other Government); ULG Wallonie (Unknown)
Responsible Party: Pr. Faiez ZANNAD, CIC-P, CHU de Nancy
Other Study IDs: 2010-A00549-30
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Cardiovascular Pathology
Keywords: nutrition; environnement; cardiovascular pathology

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urinary biological taking away: glycemia, HbA1C, insulin (specific study analyzes), total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, apolipoproteines A1 and B, numeration of blood picture, creatinin, uric acid, gamma WP, GOT, GPT, CRP; and a urinary collection (a micturition) in order to proportion the microalbuminurie. A plasmathèque will be made up, in order to measure later on biomarqueurs of the cardiovascular risk (biological collection stored with the CIC). A measurement of pollutants and poisons will be carried out starting from taking away of hair.
Oversight: Data Monitoring Committee: No

SUMMARY:
Introduction. The cardiovascular diseases, at the origin of 4 deaths out of 10, remain the leading cause of mortality in Europe. According to WHO, this tendency will spread in 2020 on a worldwide scale. These pathologies are avoidable on the whole by the adoption of healthy lifestyles. To prevent occurred of the cardiovascular affections is, more than ever, a major goal of Public health. The transborder "Great Area", localised zone in the middle of Europe between the very high cardiovascular risks of the North and the weaker risks of the South, constitutes a zone privileged for the action against the cardiovascular diseases. However, there to date does not exist any joint action in this geographical area. The Public Research centre of the Health of the Grand-Duchy of Luxembourg, the School of Public health of the University of Liege, the Clinical Center of Investigation of the University hospital of Nancy and the University hospital of the Saar wish to be linked and mutualiser their means available and their complementary competences in order to evaluate and to act on the cardiovascular health of the citizens of the "Great Area". Over one 3 years period the Nutrition project, Environment and Cardiovascular Health (NESCAV) aims at creating on the level of the Great Area a transborder alliance of prevention and promotion of cardiovascular health. This great multicentric transverse investigation and poly-set of themes will make it possible to collect relevant data on cardiovascular health of the population of the Great area.

Objective of this biomedical research project: It is about multicentric, transverse a Européenne epidemiological study aiming, through biological questionnaires and analyses, to collect information on the cardiovascular risk factors within the Great Area.

DETAILED DESCRIPTION:
Methods: In Lorraine, this study will be carried out on 800 subjects from 18 to 69 years taking part simultaneously in a quinquennial assessment of preventive medicine (CPAM), in the Centers of Preventive medicine (CMP) of Nancy and Longwy. The study will proceed on 1 year and six months, the recruitment of the volunteers will finish with the end of the year 2011. Data collected: General questionnaire, medical examination Quantification of the nutritional contributions Perception of the participant on the methods of assumption of responsibility of various risk factors cardiovascular Blood and urinary biological taking away: glycemia, HbA1C, insulin (specific study analyzes), total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, apolipoproteines A1 and B, numeration of blood picture, creatinin, uric acid, gamma WP, GOT, GPT, CRP; and a urinary collection (a micturition) in order to proportion the microalbuminurie. A plasmathèque will be made up, in order to measure later on biomarqueurs of the cardiovascular risk (biological collection stored with the CIC). A measurement of pollutants and poisons will be carried out starting from taking away of hair. (analyzes realized in Luxembourg) Data analysis: All the relative data with the participants will be anonymisées with the CMP before export to the CIC. These anonymized data will also be the subject of a treatment computerized in the countries taking part in the study, and a database common to the partners of the Great area will be made up, in order to compare the characteristics of the 3 transborder populations.

ELIGIBILITY:
Inclusion Criteria:

* men or women aged 18 till 69 years old
* living in Lorraine since 5 years
* speaking and understanding French language
* having signed the assent
* Having a social security number

Exclusion Criteria:

* taking part of the study refusal
* signature assent refusal
* pregancy
* minor people
* People under supervision or under trusteeship

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: general population
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Faiez ZANNAD, PU-PH, Principal Investigator — CIC-P
Locations (1):
- Centre médecine Preventive, Vandœuvre-lès-Nancy, France, France